CLINICAL TRIAL: NCT04837755
Title: CORONA in the Saarland
Acronym: CORSAAR
Status: Recruiting | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Robert Bals, Professor, Universität des Saarlandes
Other Study IDs: CORSAAR1
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, EDTA, PaxGene
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Cytokine measurements — The serum concentrations of multiple cytokines are measured.

SUMMARY:
The CORSAAR study is an observational, prospective study to investigate the natural biology of COVID-19

DETAILED DESCRIPTION:
Patients with all forms of COVID-19 are included and followed up. Medical history, measurements and biomarkers are registered and collected at baseline, dung hospitalization and after discharge. In addition, patients with LONG-COVID-19 are recruited.

ELIGIBILITY:
Inclusion Criteria:

all form of COVID-19 including long-COVID-19

Exclusion Criteria:

-

Ages: 0 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All COVID-19 patients in the State of Saarland
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of biomarkers with mortality and disease subgroups | 2 years after initial disease

CONTACTS AND LOCATIONS:
Locations (1):
- Saarland University, Homburg, Saarland, Germany

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol